CLINICAL TRIAL: NCT02997241
Title: Circulating Tumor DNA Predict Recurrence and Aid Treatment Decisions in Colon Cancer
Brief Title: Colon Cancer Treatment Decisions and Recurrence Predicting
Acronym: CCTDRP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: MyGenostics Inc., Beijing (Industry)
Collaborators: Chinese PLA General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: MG-WXu
Record Dates: First submitted 2016-12-13; First posted 2016-12-20 (Estimated); Last update posted 2016-12-20 (Estimated); Status verified 2016-12

CONDITIONS: Colonic Neoplasms
Keywords: Colonic Neoplasms; recurrence
MeSH Terms: conditions — Colonic Neoplasms; Recurrence | interventions — Drug Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- high genetic risk and high clinical risk (Other): on the basis of genetic risk judged by Oncocare and clinical risk judged by Clinical routine method
  Interventions: Biological: OncoCare
- low genetic risk but high clinical risk (Active Comparator): on the basis of genetic risk judged by Oncocare and clinical risk judged by Clinical routine method，randomized design，and chemotherapy for colorectal carcinoma
  Interventions: Biological: OncoCare; Drug: chemotherapy for colorectal carcinoma
- high genetic risk but low clinical risk (Active Comparator): on the basis of genetic risk judged by Oncocare and clinical risk judged by Clinical routine method
  Interventions: Biological: OncoCare; Drug: chemotherapy for colorectal carcinoma
- low genetic risk and low clinical risk (Other): on the basis of genetic risk judged by Oncocare and clinical risk judged by Clinical routine method
  Interventions: Biological: OncoCare

INTERVENTIONS:
Biological: OncoCare — Personalized monitoring
Drug: chemotherapy for colorectal carcinoma — chemotherapy for colorectal carcinoma
  Arms: high genetic risk but low clinical risk; low genetic risk but high clinical risk

SUMMARY:
The purpose of the study is to determine the relationship between change of gene copies and recurrence，and the overall survival at 5 years after chemotherapy based on clinical prognosis compared to Oncocare detection prognosis.

DETAILED DESCRIPTION:
Colorectal cancer is the third most common cancer worldwide. About two-thirds of the patients have a good therapeutic effect by combining surgical adjuvant treatment. But there are still 30-40% of patients may relapse. Efficient relapse early surveillance and accurate treatment decisions can avoid excessive medical treatment，and keep timely intervention to tumor recurrence as well. That's very important to extend the survival of patients. Currently, the efficient surveillance tools recommended by surveillance guidelines include clinical assessment, serum carcinoembryonic antigen testing, colonoscopy and CT.

Cell-free DNA(cfDNA)，the free form of DNA in the plasma，derived from the normal cells, the abnormal cells (such as tumor cells) or external (such as viral DNA). The plasma cell-free DNA derived from tumor cells is the circulating tumour DNA(ctDNA).

As most solid tumors, including CRC, release ctDNA into the blood,precision medical applications of ctDNA liquid biopsy in colorectal cancer to predict recurrence and aid treatment decisions has become a hot topic.

Recent research shows that substantially all of colorectal cancer patients have somatic genetic alterations, including both single-base mutation and larger somatic structural variations (SSVs). Mutations in these genes can be used as biomarkers to evaluate tumor burden, predict recurrence and supply information for treatment decisions through monitor and quantify ctDNA.

In this program，sequencing the tissue from colorectal cancer patients by capture technology TM and next generation sequencing(NGS),the specific somatic mutations，the so-called biomarkers, can be found.The analysis results of sequencing can help to the study of tumor molecular pathology and supply information for targetable drug.The continuous monitoring of biomarkers in the plasma can predict recurrence and supply information for treatment decisions.

In phase I trials， recruit 200 volunteers with colorectal cancer will be recruited.the investigators will test the recurrence predicting project through OncocareTM(method mentioned above). In phase Ⅱ trials，the colorectal cancer patients will be categorized into four groups on the basis of genetic risk judged by OncocareTM and clinical risk judged by Clinical routine method. Particular emphasis is on the group of low genetic risk but high clinical risk and the group of high genetic risk but low clinical risk.

The purpose of the study is to determine the relationship between change of gene copies and recurrence，and the overall survival at 5 years after chemotherapy based on clinical prognosis compared to Oncocare detection prognosis.

ELIGIBILITY:
Inclusion Criteria:

* more than eighteen, diagnosed with colorectal cancer， not chemotherapy history, Inform consent signed.

Exclusion Criteria:

* Psychosocial disorder, No inform consent signed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2017-01; Primary Completion 2017-12 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
patients treated with chemotherapy based on clinical prognosis compared to Oncocare detection prognosis | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 66 weeks

SECONDARY OUTCOMES:
the rate of gene copies change from primary detection to recurrence | From date of randomization until the date of first documented progression, assessed up to 100 weeks
Overall survival at 5 years | From date of randomization until the date of death from any cause, assessed up to 60 months

CONTACTS AND LOCATIONS:
Overall Officials: Wentong Xu, A.P., Principal Investigator — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No